CLINICAL TRIAL: NCT07294794
Title: Personalised Pharmacometabolomic-guided Strategy Trial to Optimise Treatment for Hypertension (HYPERMARKER)
Brief Title: Personalised Pharmacometabolomic-guided Strategy Trial to Optimise Treatment for Hypertension
Acronym: HYPERMARKER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other); Instituto de Investigacion Sanitaria INCLIVA (Other); University Medical Center Hamburg-Eppendorf (UKE) (Unknown); London School of Economics and Political Science (Other); Leiden University (Other); Julius Centre for Health Sciences and Primary Care, UMC Utrecht (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RG_24-123; 354889 (Other: IRAS)
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-03

CONDITIONS: Hypertension
Keywords: metabolomics; pharmacometabolomics; personalised management; blood pressure; machine learning
MeSH Terms: conditions — Hypertension | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The trial is organised into two phases. In the first phase, participants will be randomised to usual standard of care (group A) for treatment selection, or initial pharmacometabolomic approach (group B). In the second phase, participants originally randomised to group A will have their medications re-reviewed by the clinical investigator with access to the latest iteration of the pharmacometabolomic approach. Similarly, those originally randomised to group B will also potentially benefit from updates to the pharmacometabolomic approach during the course of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Up front prescription based on the usual standard of care, followed by the latest iteration of the pharmacometabolomic approach
  Interventions: Other: Standard of Care (SOC); Other: Pharmacometabolomic approach
- Group B (Experimental): Up-front initial pharmacometabolomic approach, followed by an iterated version of the pharmacometabolomic approach
  Interventions: Other: Pharmacometabolomic approach

INTERVENTIONS:
Other: Standard of Care (SOC) — Standard of care for this trial is defined according to the 2024 European Society of Cardiology Guidelines for the management of elevated blood pressure and hypertension.
  Arms: Group A
Other: Pharmacometabolomic approach — The intervention will combine metabolomic and clinical data using machine learning to provide additional information clinical investigators may utilise in their choice of blood pressure-lowering medication class for individual patients (pharmacometabolomic approach). To allow for an improved approach in the second phase of the trial, the pharmacometabolomic approach will be iterated and refined during the trial as additional metabolomic and clinical data are obtained.

SUMMARY:
High blood pressure (hypertension) affects 1 in 3 adults and can lead to serious health issues like strokes and heart attacks. Medication can lower blood pressure (BP) and reduce complications. Choosing the right medication can be challenging, potentially leading to side effects or poor control.

HYPERMARKER is testing whether providing doctors with additional information when they make a blood pressure prescription choice can improve a patient's overall blood pressure management. This includes relevant clinical information and personalised results from blood tests, brought together using computer programs (machine learning)- 'smart approach'. The blood tests check for small substances naturally produced by the body called metabolites

Developed with patient and public involvement, this proof-of-concept clinical trial will recruit 400 people across four sites in the UK, Spain, the Netherlands, and Germany. Participants must have a recent high blood pressure reading with a clinical need for medication. After providing written consent, they will provide a blood sample (to measure their metabolites) and receive a BP monitor connected to a smartphone app allowing them to measure and record their BP at home throughout the trial.

The study's main outcome is home BP readings. Participants will also complete web-based questionnaires about their health, diet, treatment experience, and healthcare usage.

Participants will be randomly assigned to two groups. Group A will receive medication based on standard clinical practice up-front, then investigators will receive output from the smart approach to refine the choice of treatment. In Group B, investigators will receive the output from the 'smart approach' initially, with further updates provided later.

Only medications licensed for hypertension will be used. All prescriptions are determined by clinicians throughout the trial.

The trial lasts 9-16 weeks. At the end, participants and their usual doctor get a copy of their BP readings and medication to guide their long-term care.

DETAILED DESCRIPTION:
Trial design and setting:

HYPERMARKER is a proof-of-concept, pragmatic, adaptive, open-label strategy trial embedded in routine clinical practice with stratified individual patient randomisation. The setting is secondary care, including four hospital sites in four countries (Germany, the Netherlands, Spain and the United Kingdom). Potential participants can be identified at sites from referrals, hospital clinics, ambulatory care centres, during hospital admissions by their care team or members of the research team contracted at the site. Eligibility should be confirmed by medically-qualified personnel. Except for the enrolment process and optional final blood test, the trial can be managed remotely, or with in-person visits as preferred by sites and participants.

The intervention will combine metabolomic and clinical data using machine learning to provide additional information clinical investigators may utilise in their choice of blood pressure-lowering medication class for individual patients (pharmacometabolomic approach). The trial is organised into two phases to iterate and improve the pharmacometabolomic approach, and ensure that all patients included in the trial have access to the intervention. In the first phase, participants will be randomised to usual standard of care (group A) for treatment selection, or initial pharmacometabolomic approach (group B). In the second phase, participants originally randomised to group A will have their medications re-reviewed by the clinical investigator with access to the latest iteration of the pharmacometabolomic approach. Similarly, those originally randomised to group B will also potentially benefit from updates to the pharmacometabolomic approach during the course of the trial.

The range of drugs considered by the pharmacometabolomic approach are well-established hypertension medications that are the core basis of usual standard of care for hypertension treatment. All prescription decisions are made by the local Investigator who should be clinically-qualified with a license to practice and prescribe.

Enrolment:

HYPERMARKER is a pragmatic clinical trial, and patients will be recruited by opportunity within the recruitment period for each site. After written informed consent, the participant will be randomised and a blood sample collected to assess their metabolomic profile. Patient demographics, medical and medication history, comorbidity burden and patient-reported outcomes are collected. The study team will set up the home blood pressure monitoring device, demonstrate to the participant, and connect it to their own mobile device. Each participant will be asked to capture at least one week of home blood pressure measurements following randomisation. Patients, clinicians and study researchers will be able to access blood pressure values and trends using the secure online trial portal.

Randomisation and treatment allocation:

Timing: Participants can only be randomised after all eligibility criteria have been confirmed and informed consent is documented.

Process: Randomisation will be stratified by site (four sites), participant age (18-69 & ≥70 years), and baseline SBP (SBP 140-159mmHg or ≥160mmHg), allocating the participants 1:1 to either Group A (initial standard of care) or Group B (up-front pharmacometabolomic approach). Investigators will randomise participants directly through the online trial platform using the Research Electronic Data Capture (REDCap) system.

Concealment of allocation: As an open-label trial, both the Investigator and participant will be aware of the allocation after randomisation, with the Investigator responsible for informing the participant about the randomised allocation.

Procedure where a participant withdraws from the trial: If a participant withdraws then their randomisation code cannot be reused. If a participant withdraws, they can be replaced.

Follow-up:

Group A Any changes or additional medication(s) will be initiated by the Investigator after the participant has completed at least one week of home blood pressure measurements. Choice of therapy will be left to the Investigator based on their usual clinical approach, and without the additional pharmacometabolomic information. Four weeks of blood pressure readings, and patient reported outcomes (PROs) completion will be requested of each participant. In the second phase, investigators are provided with the output from the latest iteration of the pharmacometabolomic approach when making their own clinical decision on what medication to prescribe. The participant is then requested to complete a further 4-weeks of blood pressure readings, and PRO completion regardless of any therapy change.

Group B The output from the pharmacometabolomic approach will be communicated within a 4-6 week period to investigators. Clinical staff will then be expected to prescribe therapy of their own choosing, ideally aligning with the pharmacometabolomic approach if deemed clinically appropriate. Four weeks of blood pressure measurements, and PRO completion will be requested of each participant. In the second phase, Clinical Investigators will receive an update from the latest iteration of the pharmacometabolomic approach and may choose to change the prescribed medication if clinically appropriate. A further 4-weeks of blood pressure measurements as well as PRO completion will be requested of participants requested regardless of any therapy change.

Blood pressure monitoring:

Participants will be requested to complete at least 3 days of blood pressure measurements at home per monitoring week. Each day consists of two readings in the morning and in the evening. Participants will receive notifications via the study app as they move through monitoring periods and by way of reminder to ensure readings are collected.

Patient Reported outcomes questionnaires:

Questionnaires can be sent by text message or email invitation and completed on a web-browser hosted by the online trial platform system - REDCap using any electronic device/system (Phone, tablet, laptop or desktop PC). Participants receive programmed reminders to complete the questionnaires.

The following questionnaires will be collected:

Quality of life: The EuroQOL EQ-5D-5L questionnaire will be collected at baseline, and following each phase of the trial.

Healthcare resource utilisation: This questionnaire collects data relevant to direct and indirect healthcare utilisation and will be collected at baseline, and following each phase of the trial.

Adherence questionnaire: Participants will be asked about whether they are taking the suggested anti-hypertensive medication and if they have any perceived adverse reactions. It will be collected following each phase of the trial. Socioeconomic & Demographic questionnaire. This questionnaire will be optional for participants and sent at baseline.

Dietary intake: A dietary intake questionnaire will be completed by participants at site using an electronic device/system (Phone, tablet, laptop or desktop PC). Questionnaires will be hosted by myfood24 (Dietary Assessment Ltd), for sites in the UK and collect data regarding participants food and drink consumption from the previous 24hrs.

End of trial:

Each participant will be asked to attend their local research site to have an optional blood sample to assess changes in their metabolomic profile; this is for research purposes only and will not contribute to clinical care. The end of study for each participant is defined as the date of the last patient-reported blood pressure or patient-reported outcome.

Public and Patient Involvement in the study design and methodology:

A patient and public involvement (PPI) group with representatives from all four trial site countries have reviewed the trial design and content of key trial documents such as the protocol, participant information leaflet, participant information video and the informed consent form. The PPI group have also tested the at home blood pressure device and mobile application as well as patient-reported outcome questionnaires. Changes including to the content, delivery platform and design have been made following PPI feedback to ensure participants will understand and accept what will happen to them in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Systolic blood pressure ≥140 mmHg on any blood pressure recording method (office, home or ambulatory)
2. Age 18 years or older
3. Clinical indication for antihypertensive therapy

Exclusion Criteria:

1. Systolic blood pressure ≥180 mmHg on any blood pressure recording method (office, home or ambulatory)
2. Potential secondary cause of hypertension, including but not limited to renovascular hypertension, endocrine conditions, chronic kidney disease, coarctation of the aorta or medication related.
3. Three or more current anti-hypertensive medications
4. Planned intervention for hypertension, such as renal denervation
5. Severe kidney disease (estimated glomerular filtration rate <30 mL/min)
6. Diagnosis of known heart failure with left ventricular ejection fraction <40%
7. Stroke or myocardial infarction within the last 6 months
8. Pregnancy, planning for pregnancy, or breastfeeding
9. Participant whom the Clinical Investigator deems otherwise ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in home Systolic Blood Pressure | 5 weeks
  Change in home SBP will be derived from all available patient-measured SBP recordings in the study smartphone application, comparing the intervention and standard of care groups at the end of the first phase of the trial. This includes 1-week of monitoring after enrolment (anticipated minimum of 12 recordings) and at least 4-weeks of monitoring after therapy change (anticipated minimum of 48 recordings).

SECONDARY OUTCOMES:
Proportion of participants achieving a target home SBP of 120-129mmHg using the average of the final 3 days of blood pressure measurements. | 4 weeks
  Comparing the intervention and standard of care groups at the end of the first phase of the trial
Proportion of participants reporting any treatment-related adverse effects compiled from the Summary of Product Characteristics from the different classes of anti-hypertensive medications | 4 weeks
  Comparing the intervention and standard of care groups at the end of the first phase of the trial
Proportion of participants reporting withdrawal of an anti-hypertensive medication. | 4 weeks
  Comparing the intervention and standard of care groups at the end of the first phase of the trial
Proportion of participants reporting ≥90% adherence to prescribed anti-hypertensive medication | 4 weeks
  Comparing the intervention and standard of care groups at the end of the first phase of the trial
Rate of change in home SBP using all available SBP measurements, averaged per week. | 5 weeks
  Comparing the intervention and standard of care groups at the end of the first phase of the trial
Change in home diastolic blood pressure derived from all available blood pressure recordings. | 5 weeks
  Comparing the intervention and standard of care groups at the end of the first phase of the trial
Change in home SBP using all available SBP measurements. | 9 weeks
  Comparing the iterated pharmacometabolomic approach versus the initial pharmacometabolomic approach, and the iterated pharmacometabolomic approach versus initial standard of care
Patient-reported treatment-related side effects | 8 weeks
  Comparing the iterated pharmacometabolomic approach versus the initial pharmacometabolomic approach, and the iterated pharmacometabolomic approach versus initial standard of care
Proportion and number of serious adverse events, including all-cause hospitalisation and death | 9 weeks
  Comparing any pharmacometabolomic approach versus standard of care
Proportion and number of healthcare utilisation events, including details on hospitalisation (frequency, cause, type [outpatient, emergency, admission] and length of stay) and primary care interaction (frequency, cause and type [doctor, nurse, other | 9 weeks
  Comparing any pharmacometabolomic approach versus standard of care
Patient-reported quality of life using the EQ-5D-5L summary index score and visual analogue scale. | 9 weeks
  Comparing any pharmacometabolomic approach versus standard of care

OTHER OUTCOMES:
Change in metabolomic profile from baseline to (optional) follow-up blood sample, stratified by class of anti-hypertensive medication (exploratory). | 9weeks
  This outcome is unrelated to the randomised group
Association between dietary intake, metabolomic profile and blood pressure response to prescribed antihypertensive treatment (exploratory). | 9 weeks
  Outcome is unrelated to the randomised group
Life years and quality-adjusted life year (QALY) gained | 9 weeks
Net monetary benefits of the pharmacometabolomic approach | 9 weeks
Difference in healthcare utilisation and cost estimates between standard care and the pharmacometabolomic approach | 9 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- University Medical Centre Utrecht, Utrecht, Netherlands
- INCLIVA, Biomedical Research Institute, Valencia, Spain
- University Hospitals Birmingham, NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No